CLINICAL TRIAL: NCT03418506
Title: Knowledge and Awareness Regarding Association of Arecanut/Betel Quid and With Oral Cancer and Other Serious Illnesses Among Children 11-16 Years; A Cluster Randomized Intervention Study
Brief Title: Improvement in Knowledge and Perception About Hazards of Smokeless Tobacco
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aga Khan University (Other)
Collaborators: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, Shafquat Rozi, Assistant Professor, Aga Khan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB-756DUHS/approval/2016/310
Record Dates: First submitted 2018-01-17; First posted 2018-02-01 (Actual); Last update posted 2018-02-05 (Actual); Status verified 2018-02

CONDITIONS: Smokeless Tobacco Cessation
Keywords: Smokeless tobacco; adolescent; oral cancer; betal quid; areca nut
MeSH Terms: conditions — Tobacco Use Cessation; Tobacco Use; Mouth Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): A SMOKELESS TOBACCO AWARENESS PROGRAM was conducted for 2 consecutive weeks in all the selected schools. The intervention programme comprised of health education sessions that emphasized on the hazard of betel quid, areca-nut and smokeless tobacco. The sessions included 30 minutes power point presentation, posters, one pictorial booklets on the hazards of use of various tobacco products. Moreover we played a 30 minutes game show at follow-up visit. After completion of 2 weeks intervention programme, the same group of students completed the post-test questionnaire. Educational materials about hazards of betel quid, areca-nut and smokeless tobacco were distributed to both intervention and control groups.
  Interventions: Behavioral: SMOKELESS TOBACCO AWARENESS PROGRAM
- Control (No Intervention): No specific education will be given to the control group.

INTERVENTIONS:
Behavioral: SMOKELESS TOBACCO AWARENESS PROGRAM — A SMOKELESS TOBACCO AWARENESS PROGRAM was conducted for 2 consecutive weeks in all the selected schools. The intervention programme comprised of health education sessions that emphasized on the hazard of betel quid, areca-nut and smokeless tobacco. The sessions included 30 minutes power point presentation, posters, one pictorial booklets on the hazards of use of various tobacco products. Moreover we played a 30 minutes game show at follow-up visit. After completion of 2 weeks intervention programme, the same group of students completed the post-test questionnaire. Educational materials about hazards of betel quid, areca-nut and smokeless tobacco were distributed to both intervention and control groups.
  Arms: Intervention

SUMMARY:
Oral cancer is a serious and growing problem in many parts of the globe. Oral cancer is the eighth most common cancer worldwide.The annual estimated incidence is around 275,000 for oral and 130,300 for pharyngeal cancers excluding nasopharynx, two-thirds of these cases occurring in developing countries. In Pakistan, it is the second most common cancer in women and third most common cancer in men. The Age Standardized Rates (ASR) for oral cancers are 13.8 and 14.1 in males and females respectively.To the best of investigators knowledge, no intervention study has been done to improve knowledge and awareness of adults regarding association of areca nut/betel quid with oral cancer. Therefore, the study aims to implement a cluster randomized intervention trial in secondary schools to improve the knowledge and awareness regarding this association among children 11-16 years. For resource poor countries such as Pakistan, it is imperative to prevent oral cancer by improving knowledge about its important risk factor such as betel quid, areca nut and chew tobacco. A school-based intervention study will be carried out in secondary schools in Karachi. The target population will be male and female school students in school grades 6 to 10 with intervention group and control group at each site. School-based educational intervention will be given to the intervention group while no specific education will be given to the control group. Differences in attitudes, knowledge and behaviors between the intervention and control groups will be compared each site separately before and after the intervention. The minimum sample size required was 22 schools (clusters). The number of subjects in each arm will be 529 with average cluster size of 50. The selected schools will be randomly assigned to a control group or Interventions group. Randomization will be done at the school level to avoid contamination between groups.The health education programme will be conducted for 3 consecutive weeks in one academic year for all the selected schools.

DETAILED DESCRIPTION:
Oral cancer is a serious and growing problem in many parts of the globe. Oral cancer is the eighth most common cancer worldwide. There is a wide geographical variation (approximately 20-fold) in the incidence of this cancer. In South and South East Asia, 40% of the people with cancers have been diagnosed with it. Age-adjusted rates of oral cancer in India is high, that is, 20 per 100,000 population and accounts for over 30% of all cancers in the country. In Pakistan, it is the second most common cancer in women and third most common cancer in men.The Age Standardized Rates (ASR) for oral cancers are 13.8 and 14.1 in males and females respectively. Smoking, alcohol consumption and sunlight have been implicated in the development of oral cancers in the developed countries. In addition to these, developing countries have their own set of risk factors.These include poor infrastructure of the health care system, illiteracy, poor socioeconomic status. A common risk factor shared by populations from all over the world is substance abuse.There exists a large volume of literature which links betel nut, areca, chewable tobacco and tobacco with development of cancer.

A study from South Asia have reported the risk of oral cancer and the use of oral tobacco in various forms including ''paan'' with and without tobacco. A case-control study from Thailand reported that, among all components of the betel quid, the presence in the quid of red slaked lime had the strongest effect on the risk of oral cancer (OR,10.67; 95% CI = 2.27-50.08). A recently published meta-analysis also explores the relationship between betel quid chewing and risk of oral and oropharyngeal cancers.

Oral diseases are a major global health burden despite considerable investment in research and dental services. A meta-analysis of fifteen case control studies (4,648 cases; 7,847 controls) has shown betel quid to have an independent positive association with oral cancer, with OR = 2.82 (95% CI = 2.35-3.40). Studies conducted in Pakistan report about knowledge, perception and correlation of betel quid and head and neck cancer.

The study aims to implement a cluster randomized intervention trial in secondary schools to improve the knowledge and awareness regarding this association among children 6-10 years. For resource poor countries such as Pakistan, it is imperative to prevent oral cancer by improving knowledge about its important risk factor such as betel quid, areca nut and chew tobacco.

Methods:

Study Design and Setting:

A school-based intervention study will be carried out in secondary schools in Karachi. The target population will be male and female school students in school grades 6 to 10 with intervention group and control group at each site.

Sample Size:

Sample size was calculated using the computer program WHO ACluster. The minimum sample size required is 22 schools (clusters) with 95% confidence interval, 80% power, and ICC= 0.2. The difference to be detected was 2 with standard deviation 9.5. The number of subjects in each arm will be 529 with average cluster size of 50.

Sampling:

A two-stage cluster sampling with stratification based on school type (government or private) will be employed. A multistage cluster sampling with stratification on school type (government or private) will be employed for the selection of schools and recruitment of adolescents. After stratification schools will be selected randomly proportionate to the number of type of school from district east of Karachi. Each school will be considered as a cluster. Schools will be the primary unit of randomization. Recruitment of participating schools will be based on the willingness to participate in the study. One class will be selected randomly from each of selected secondary (grades 6-10) schools and all the students in the selected classes will be invited to participate in the survey. Hence, equal number of clusters will be selected in both groups.

Randomization:

The selected schools will be randomly assigned to a control group or Interventions group. Randomization will be done at the school level to avoid contamination between groups.

Study procedure:

Approval for the design and data collection procedures was obtained beforehand from the ethics committee of the School. An approval was obtained from school authority after explaining the purpose of the study. Written informed consent was taken from all participating schools and it will be communicated to the students that participation is completely voluntary. Absolute confidentiality of the data will be maintained throughout the study.

School-based educational intervention will be given to the intervention group while no specific education will be given to the control group. Pre and post-test questionnaires will be administered one week before and one week after the program intervention, respectively. Tests will be administered in the students' usual classroom by research assistants under the supervision of the researchers who are not affiliated with the schools.

Intervention Programme:

The health education programme will be conducted for 2 consecutive weeks in one academic year for all the selected schools. The intervention programme will comprise of health education sessions that will emphasize on the hazard of betel quid and areca nut and chew tobacco. This will be conducted through posters, pictorial booklets, video shows, and short documentaries on the hazards of use of various tobacco products. The programme will be conducted by a trained team. Educational materials about hazards of betel quid and areca nut will be distributed to both intervention and control groups.

Training sessions:

The programme will be conducted by a professional team of physicians trained in this field. A one-day training session for the program providers will be designed to maximize the success of the program implementation.

Plan of Analysis:

Investigators will perform analysis using STATA version 12. Descriptive statistics will be computed for categorical variables by computing their frequencies & assessed by chi square. The distribution of quantitative variables will be computed by their means and standard deviations & assessed by independent t test or median with inter-quartile range (IQR) depending on distribution of the variables. Investigators will perform multivariable analysis using generalizing estimating equation (GEE) to consider the clustering structure of the data. Crude odds ratio (OR) and their 95% confidence interval (CI) will be calculated using univariate GEE. All the variables with a p-value of less than 25% significance will be selected for inclusion in the multivariable analysis.

Confounding will be assessed by change in estimate of coefficient by 15%. After developing main effect model, significance of all biologically plausible interactions will be evaluated for inclusion in multivariable model.

Interim analysis:

Interim analysis will be conducted, if required, after completion of 50% of the follow-ups to see the effect of educational intervention programme on the participant's knowledge.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for cluster/school

  * High schools registered with Board of Secondary Education Karachi
  * The schools should have at least 15 students in each grade.
  * School authorities grant permission to conduct the research study in their school.

Inclusion criteria (For individual)

* Both Male/ female students from grades 6-10.
* Resident of selected areas where the schools are located for at least one year.

Exclusion Criteria:

-

Ages: 11 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1327 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2017-11-30 (Actual)

PRIMARY OUTCOMES:
Knowledge about hazards of smokeless tobacco | 6 months
  Knowledge about hazards of smokeless tobacco will be measured by a validated questionnaire from male and female school students studying in grades 6 to 10.

SECONDARY OUTCOMES:
Attitude about hazards of smokeless tobacco | 6 months
  Attitude about hazards of smokeless tobacco will be measured by a validated questionnaire from male and female school students studying in grades 6 to 10.
Perception about hazards of smokeless tobacco | 6 months
  Perception about hazards of smokeless tobacco will be measured by a validated questionnaire from male and female school students studying in grades 6 to 10.

CONTACTS AND LOCATIONS:
Overall Officials: Zahid Butt, PhD, Study Director — British Columbia
Locations (1):
- Aga Khan University, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No
It will depend on the requirement of the journal

REFERENCES:
- [Derived] Rozi S, Zahid N, Roome T, Lakhdir MPA, Sawani S, Razzak A, Butt ZA. Effectiveness of a School Based Smokeless Tobacco Intervention: A Cluster Randomized Trial. J Community Health. 2019 Dec;44(6):1098-1110. doi: 10.1007/s10900-019-00689-8. PMID 31267293